## Collaborative-Care Rehabilitation to Improve Functional Outcomes after Dysvascular Amputation

Statistical Analysis Plan Version Date: 01.05.2014

Between-group differences in all outcomes at 12- and 24-week tests will be evaluated using maximum likelihood estimation in a multivariate repeated measures model. The maximum likelihood method uses all available data and provides unbiased estimates under the assumption that missing data are missing at random. The model for each outcome will be controlled for baseline value of the outcome, rehabilitation clinic site (VA/non-VA), diagnosis of DM, and diagnosis of PAD. Estimated group means and within-group mean changes over time for each outcome will be reported with 95% confidence intervals. This early phase study is powered for one endpoint; multiple secondary endpoints are reported to guide further research without adjustment for multiplicity.